CLINICAL TRIAL: NCT02775617
Title: Impact of Combined Azithromycin and Ivermectin Mass Drug Administration for Yaws and Scabies - Impact on Impetigo and Skin Microbiology
Brief Title: Azithromycin - Ivermectin Mass Drug Administration for Skin Disease
Acronym: AIM-Skin
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Collaborators: Atoifi Adventist Hospital, Solomon Islands (Unknown); Kirby Institute (Other Government); Murdoch Childrens Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 35148A
Record Dates: First submitted 2016-02-24; First posted 2016-05-17 (Estimated); Results first posted 2019-09-13 (Actual); Last update posted 2019-09-17 (Actual); Status verified 2019-09

CONDITIONS: Scabies; Yaws; Impetigo
MeSH Terms: conditions — Scabies; Yaws; Impetigo | interventions — Ivermectin; Azithromycin; Permethrin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Parallel Treatment (Other): Site 1- Parallel Treatment Arm Single dose azithromycin (for yaws) and Ivermectin/Permethrin (for scabies) will be offered on D1. A second dose of Ivermectin/Permethrin will be offered 7-14 days later.
  Interventions: Drug: Ivermectin; Drug: Azithromycin; Drug: Permethrin
- Sequential Treatment (Other): Site 2- Serial Treatment Arm Ivermectin/Permethrin (for scabies) will be offered on D1 with a second dose of Ivermectin/Permethrin offered 7-14 days later..
  Single dose azithromycin (for yaws) will be offered at the twelve month follow-up visit.
  Interventions: Drug: Ivermectin; Drug: Azithromycin; Drug: Permethrin

INTERVENTIONS:
Drug: Ivermectin — Participants will be offered treatment for both yaws and scabies either in parallel or in sequence. Ivermectin will be offered as a a single dose 200μg/kg on Day 1 and Day 8.
Drug: Azithromycin — Participants will be offered treatment for both yaws and scabies either in parallel or in sequence. Azithromycin will be offered as single dose of 30mg/kg, max 2G.
Drug: Permethrin — Participants will be offered treatment for both yaws and scabies either in parallel or in sequence. Individuals with a contra-indication to ivermectin will be offered Permethrin instead.

SUMMARY:
This is an open-label prospective community intervention trial to assess the impact of community mass treatment with azithromycin for yaws and ivermectin for scabies, on non-yaws bacterial skin infections.

Communities will be randomised to receive standard treatment for both yaws and scabies either in parallel (site 1) or in sequence (site 2).

Treatment of yaws:

Single dose of Azithromycin (30mg/kg, max 2G).

Treatment of scabies:

Either an oral dose of Ivermectin (200μg/kg) or permethrin cream for those with a contraindication to Ivermectin (WT<15kg, pregnant or breastfeeding women) given in 2 doses 7-14 days apart.

Investigators will complete a clinical and microbiological assessment of bacterial skin disease at baseline and at 12 months to assess the impact of treatment on the prevalence of bacterial infection and the emergence of antimicrobial resistance.

Primary Outcome

1. Difference in the change in prevalence of impetigo between baseline and 12- months between the parallel and the sequential treatment arms.

   Secondary Outcomes
2. Change in the proportion of swab samples from which S. pyogenes is cultured between baseline and follow-up in the two arms
3. The proportion of samples from which a drug-resistant isolate of S.pyogenes is cultured in the two arms

ELIGIBILITY:
Inclusion Criteria:

* All community members are able to be included in the study.

Exclusion Criteria:

* Allergy to any of the components of the allocated drug regimen

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1291 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2018-02-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Marks, Principal Investigator — London School of Hygiene and Tropical Medicine
Locations (1):
- Atoifi Adventist Hospital, Atoifi, Malaita Province, Solomon Islands

IPD SHARING:
Plan to Share IPD: Undecided
Anonymised data may be made available

REFERENCES:
- [Derived] Marks M, Toloka H, Baker C, Kositz C, Asugeni J, Puiahi E, Asugeni R, Azzopardi K, Diau J, Kaldor JM, Romani L, Redman-MacLaren M, MacLaren D, Solomon AW, Mabey DCW, Steer AC. Randomized Trial of Community Treatment With Azithromycin and Ivermectin Mass Drug Administration for Control of Scabies and Impetigo. Clin Infect Dis. 2019 Mar 5;68(6):927-933. doi: 10.1093/cid/ciy574. PMID 29985978

RESULTS

PARTICIPANT FLOW:
Groups:
- Sequential Treatment: Site 2- Serial Treatment Arm Ivermectin/Permethrin (for scabies) will be offered on D1 with a second dose of Ivermectin/Permethrin offered 7-14 days later..
  Single dose azithromycin (for yaws) will be offered at the twelve month follow-up visit.
  Ivermectin: Participants will be offered treatment for both yaws and scabies either in parallel or in sequence. Ivermectin will be offered as a a single dose 200μg/kg on Day 1 and Day 8.
  Azithromycin: Participants will be offered treatment for both yaws and scabies either in parallel or in sequence. Azithromycin will be offered as single dose of 30mg/kg, max 2G.
  Permethrin: Participants will be offered treatment for both yaws and scabies either in parallel or in sequence. Individuals with a contra-indication to ivermectin will be offered Permethrin instead.
Period: Overall Study
Arm/Group | Parallel Treatment | Sequential Treatment
Started | 653 (Participants are seen at via a survey of the community. 92.6% of the resident population) | 638 (Participants are seen at via a survey of the community. 88.9% of the resident population)
Completed | 605 (Participants are seen at via a survey of the community. 96.3% of the resident population) | 478 (Participants are seen at via a survey of the community. 76.2% of the resident population)
Not Completed | 48 | 160

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Parallel Treatment | Sequential Treatment | Total
Number analyzed (Participants) | 653 | 638 | 1291
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 24 [10 to 45] | 25 [12 to 47] | 25 [10 to 47]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 335 | 312 | 647
  Male | 318 | 326 | 644
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 653 | 638 | 1291
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Solomon Islands | 653 | 638 | 1291

OUTCOME MEASURES:

1. Primary Outcome: Impetigo Prevalence at 12 Months
Description: Change in prevalence of impetigo between baseline and 12-months
Time Frame: Baseline and 12 months
Population: At the baseline survey 653 individuals were seen in the Parallel arm and 638 in the sequential treatment arm.
  At the 12 month survey 605 individuals were seen in the Parallel arm and 478 in the sequential treatment arm
Measure: Number; unit: Cases of impetigo
Arm/Group | Parallel Treatment | Sequential Treatment
Number analyzed (Participants) | 653 | 638
Cases of impetigo
  Cases Impetigo at Baseline | 79 | 66
  Cases Impetigo at 12 Months: number analyzed (Participants) | 605 | 478
  Cases Impetigo at 12 Months | 20 | 12

2. Secondary Outcome: Group A Streptococcus at 12 Months
Description: Change in the percentage of swab samples from which S. pyogenes is cultured between baseline and 12 month follow-up in the two arms
Time Frame: 12 Months
Population: Samples were collected at twelve months from individuals with clinical impetigo and cultured for both pyogenic streptococci and S.aureus.
  This analysis is therefore restricted to the subset of patients who had impetigo from which a swab was collected
Measure: Number; unit: Change in number swabs with S.pyogenes
Arm/Group | Parallel Treatment | Sequential Treatment
Number analyzed (Participants) | 54 | 41
Change in number swabs with S.pyogenes
  Swabs containing S.pyogenes at baseline: number analyzed (Participants) | 38 | 35
  Swabs containing S.pyogenes at baseline | 17 | 28
  Swabs containing S.pyogenes at 12 months: number analyzed (Participants) | 16 | 6
  Swabs containing S.pyogenes at 12 months | 4 | 1

3. Secondary Outcome: Antimicrobial Resistance in Culture Isolates
Description: The proportion of samples from which a drug-resistant isolate of S.pyogenes is cultured in the two arms
Time Frame: 12 Months
Population: This analysis was restricted to the subset of patients in whom S.pyogenes was isolated on a swab
Measure: Number; unit: Number of swabs
Arm/Group | Parallel Treatment | Sequential Treatment
Number analyzed (Participants) | 33 | 34
Number of swabs
  % Swabs with resistance at baseline: number analyzed (Participants) | 17 | 28
  % Swabs with resistance at baseline | 0 | 0
  % Swabs with resistance at 12 months: number analyzed (Participants) | 16 | 6
  % Swabs with resistance at 12 months | 0 | 0

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Parallel Treatment | Sequential Treatment
All-Cause Mortality (participants affected / at risk) | 0/653 | 0/638
Serious Adverse Events (participants affected / at risk) | 0/653 | 0/638
Other Adverse Events (participants affected / at risk) | 0/653 | 0/638

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-02-17): https://cdn.clinicaltrials.gov/large-docs/17/NCT02775617/Prot_SAP_000.pdf